CLINICAL TRIAL: NCT03322475
Title: Evaluation of the Efficacy and Safety of PiQo4 for Facial Skin Rejuvenation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Focus Medical, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Focus-PiQo4 Rejuvenation-17-02
Record Dates: First submitted 2017-10-24; First posted 2017-10-26 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Skin Rejuvenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Facial skin rejuvenation (Experimental): Facial skin rejuvenation using PiQo4 laser system
  Interventions: Device: PiQo4 laser system

INTERVENTIONS:
Device: PiQo4 laser system — The PiQo4 laser system

SUMMARY:
A total of at least 20 healthy subjects at a single site, with at least two facial sub-areas with visible wrinkles with pigmentation and/or acne scars who wish to improve their skin appearance will be enrolled into the study. subjects will receive 3 treatments and return to follow-up visits at 1, 3, and 6 months following the last treatment.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be entered into the study:

* Healthy Female/Male.
* Age= 18-70 (Adults).
* Fitzpatrick skin phototype = I-V
* Exhibiting at least two facial sub-areas with visible wrinkles with pigmentation and/or acne scars.
* Able to read, understand and provide written Informed Consent.
* Able and willing to comply with the treatment/follow-up schedule and post treatment care
* Willingness to provide a brief medical history including disclosure of any prescribed or over-the-counter medications taken within the past 6 months.
* Willingness to allow Focus Medical (the study Sponsor) and Lumenis and the investigators to use de-identified photographs of the treated area for presentation and publication purposes.
* Daily use of sunscreen for the duration of the study
* Women of child-bearing potential are required to use a reliable method of birth control (such as an intrauterine device, birth control pills, condom with spermicidal, NuvaRing, partner with vasectomy, Implanon or other FDA-approved devices, or abstinence) during the course of the study.

Exclusion Criteria:

Any of the following will exclude the subject from the study:

* Pregnant, intending to become pregnant during the course of study, less than 3 months postpartum or less than 3 months after completion of breastfeeding
* Prior skin laser, light or other energy device treatment in treated area within 6 months of initial treatment or during the course of the study.
* Known hypersensitivity or contraindications to anesthetic agents including lidocaine and its derivatives, and Toradol.
* Having a history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treated area, unless treatment is conducted following a prophylactic regimen.
* History of post inflammatory pigmentary disorders, particularly a tendency for hyper- or hypo-pigmentation.
* Having Melasma.
* Having multiple dysplastic Nevi in are to be treated.
* Having an excessive underlying vascular conditions (e.g. dense network of capillaries).
* History of keloid scarring or of abnormal wound healing.
* Suffering from current or history of significant skin conditions in the treated area or inflammatory skin conditions.
* History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications.
* Having a known anticoagulative or thromboembolic condition or taking anticoagulation medications one week prior to and during the treatment course (to allow inclusion, temporary cessation of use as per the subject's physician's discretion).
* Having a neurological disorder (including Multiple Sclerosis, Parkinson's disease).
* Having seizure disorder.
* Having fibromyalgia.
* Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
* Participation in a study of another device or drug within three months prior to enrolment or during the study.
* Significant concurrent illness (e.g. uncontrolled diabetes) or any disease state that in the opinion of the Investigator would interfere with the treatment or healing process
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.
* Subjects who are opposed to possible damage to the hair follicles with possible loss of hair in the treatment area.
* Received the following treatments in the area of the face to be treated during or within the noted timeframes prior to the study treatment:

  1. Dermabrasion or chemical peel treatment within 3 months.
  2. Any devices and/or Botox treatment within 6 months.
  3. Collagen/fat injections or other methods of augmentation with injected or implanted material in the treated area within 9 months.
  4. Resurfacing procedure, face lift or eyelid surgery within a year.
  5. Having a permanent implant in the facial skin area, such as an injected chemical substance.
  6. Any other surgery in treated area within 9 months of initial treatment or during the course of the study
  7. Use of retinoids, antioxidants or therapeutic skin nourishing supplements at medicinal concentration within 2 months and oral retinoids within 6 months of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-03-12 (Actual); Primary Completion 2019-07-30 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Fitzpatrick Elastosis Score (FES) scale | Baseline, 1 month follow up
  Fine lines/wrinkles and elastosis improvement will be classified by the Fitzpatrick-Goldman Elastosis and Wrinkles scales: Class I, Class II or Class III.
Overall Global Aesthetic Improvement (GAI) Scale | Baseline, 1 month follow up
  The global aesthetic improvement (GAI) scale will be used by the investigator to grade improvement in the following categories: 1) Fine lines/wrinkles; 2) texture 3) Pigmentation 4) Acne scars. Score 0-Worse, Score 1-No Change, Score 2- Somewhat improved, Score 3- Moderately improved, Score 4-Very Much Improved.

SECONDARY OUTCOMES:
Fitzpatrick Elastosis Score (FES) scale | Baseline, 3 month follow up
  Skin improvement on the FES scale will be classified by the Fitzpatrick-Goldman Elastosis and Wrinkles scales at the 3 month-follow-up visits as compared to baseline.
  Classification: Class I, Class II or Class III.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Ross, MD, Principal Investigator — Scripps Clinic Carmel Valley
Locations (1):
- Scripps Clinical Research Services, La Jolla, California, United States